CLINICAL TRIAL: NCT07210359
Title: Evaluation of Regenerative Endodontic Treatment for Immature Teeth Using Two Different Forms of Demineralized Dentin Matrix and RetroMTA: Randomized Controlled Clinical Trial
Brief Title: Evaluation of Regenerative Endodontic Treatment for Immature Teeth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hisham Mahmoud Hamdy Abada, lecturer at Endodontic department, Kafrelsheikh University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 663
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Pulpal Necrosis
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Demineralized Dentin Matrix

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- treated hyman dentin matrix hydrogel (Active Comparator): material used for regenerative dentistry
  Interventions: Procedure: Theracal LC - Demineralized dentin matrix combination; Procedure: Retro Mta
- Theracal LC- Demineralized dentina matrix combination (Active Comparator): material used for regenerative dentistry
  Interventions: Procedure: human treated dentin matrix hydrogel; Procedure: Retro Mta
- RetroMTA (Active Comparator): material used for regenerative dentistry
  Interventions: Procedure: human treated dentin matrix hydrogel; Procedure: Theracal LC - Demineralized dentin matrix combination

INTERVENTIONS:
Procedure: human treated dentin matrix hydrogel — material used for regenerative dentistry
  Other Names: demineralized dentin matrix
  Arms: RetroMTA; Theracal LC- Demineralized dentina matrix combination
Procedure: Theracal LC - Demineralized dentin matrix combination — material used for regenerative dentistry
  Arms: RetroMTA; treated hyman dentin matrix hydrogel
Procedure: Retro Mta — material used for regenerative dentistry
  Arms: Theracal LC- Demineralized dentina matrix combination; treated hyman dentin matrix hydrogel

SUMMARY:
The goal of this clinical trial is to evaluate if regenerative endodontic treatment using two different forms of demineralized dentin matrix (DDM) can effectively treat immature permanent single-rooted teeth compared to treatment using RetroMTA in patients aged 9 to 15 years. The main questions it aims to answer are:

Does the use of DDM improve clinical and radiographic outcomes such as root length, dentinal wall thickness, and apex closure?

Is DDM a viable bioactive alternative to RetroMTA as a coronal sealing material in regenerative endodontic procedures?

Researchers will compare three groups: one using RetroMTA, one using a DDM-TheraCal LC mixture, and one using TDM-Hydrogel, to see if these materials differ in their effects on regenerative outcomes.

Participants will:

Undergo two treatment visits including canal disinfection, induction of bleeding to form a blood clot scaffold,

Receive placement of one of the study materials over the blood clot as a coronal barrier,

Have clinical examinations and CBCT imaging at baseline and multiple follow-ups up to 12 months to assess treatment success through signs, symptoms, and radiographic changes.

DETAILED DESCRIPTION:
The study was conducted as a split-mouth randomized clinical trial, approved by research ethics committee, Faculty of Dentistry, Kafrelsheikh University, and carried out at Endodontic Department, Faculty of Dentistry, Kafrelsheikh University. 36 patients of both sexes aged from 9 to 15 years old were selected with an immature teeth with teeth diagnosed as either vital (asymptomatic irreversible pulpitis or symptomatic irreversible pulpitis and the bleeding didn't stop after 5 minutes application of hemostatic agent) or non-vital pulp are indicated for regenerative endodontic procedure.

Patients will be divided randomly into three equal groups (n = 12):

Group 1(control group): Revascularization will be done using blood clot and RetroMTA as coronal barrier.

Group 2: Revascularization will be done using blood clot and DDM-TheraCal LC mixture paste as coronal barrier.

Group 3: Revascularization will be done using blood clot and TDM-Hydrogel as coronal barrier.

CBCT image will be obtained for baseline records before treatment and after placement of the final resin restoration, then the patients will be recalled after 3, 6, 9 and 12 months for evaluating any changes in dentin bridge formation, root length, root canal width, apex diameter and lesion size if present.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients (i.e., free of any systemic diseases).
* Patients presenting with immature permanent single-rooted teeth.
* Age: 9 -15 years.
* Teeth diagnosed as either vital (asymptomatic irreversible pulpitis or symptomatic irreversible pulpitis and the bleeding didn't stop after 5 minutes application of hemostatic agent) or non-vital pulp.

Exclusion Criteria:

* Patients who are allergic to any drugs used in this study or with systemic illness
* Teeth that are grossly decayed or fractured and require post and core as final restorations
* Presence of periodontal pockets greater than 4 mm.
* Radiographical evidence of apical foramen less than 1 mm.
* Presence of periapical radiolucency exceeding 10 mm.
* Presence of external or internal root resorption.
* Patients with a history of major surgeries like cardiac, kidney transplantation, haemodialysis.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maturation of root | year
  root length increase, root width increase, apical formane closes and dentinal bridge formation over regenerated pulp

SECONDARY OUTCOMES:
resolve of apical lesion if present | 1 year
  if there is any apical lesion, it will resolve and new bone formation takes place.

OTHER OUTCOMES:
regain sensibility of pulp | 1 t 2 years
  nerve supply of pulp is regenerated with time but not primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Abada, Doctors, Principal Investigator — Academic
Locations (1):
- KafrelsheikhU, Kafr ash Shaykh, Kafr Elsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided